CLINICAL TRIAL: NCT05158140
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of the Concomitant Administration of Either 23-Valent Pneumococcal Polysaccharide Vaccine or 15-Valent Pneumococcal Conjugate Vaccine With a Booster Dose of SARS-CoV-2 mRNA Vaccine in Healthy Adults 50 Years of Age or Older.
Brief Title: Safety, Tolerability, and Immunogenicity of V110 or V114 Co-administered With a Booster Dose of mRNA-1273 in Healthy Adults (V110-911)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V110-911
Record Dates: First submitted 2021-12-03; First posted 2021-12-15 (Actual); Results first posted 2024-02-13 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Pneumococcal Infection
MeSH Terms: conditions — Pneumococcal Infections | interventions — 2,4,5,4'-tetrachlorodiphenylsulfoxide; 23-valent pneumococcal capsular polysaccharide vaccine; Vaccines; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- V110 Concomitant with mRNA-1273 (V110 Concomitant) (Experimental): Participants received a single 0.5 mL intramuscular (IM) injection of V110 concomitantly with a single 0.25 mL IM injection of mRNA-1273 on Day 1, followed by a single 0.5 mL IM injection of placebo for V110 on Day 30.
  Interventions: Biological: V110; Biological: mRNA-1273; Biological: Placebo for V110
- V110 Nonconcomitant with mRNA-1273 (V110 Nonconcomitant) (Experimental): Participants received a single 0.5 mL IM injection of placebo for V110 on Day 1 concomitantly with a single 0.25 mL IM injection of mRNA-1273, followed by a single 0.5 mL IM injection of V110 on Day 30.
  Interventions: Biological: V110; Biological: mRNA-1273; Biological: Placebo for V110
- V114 Concomitant with mRNA-1273 (V114 Concomitant) (Experimental): Participants received a single 0.5 mL IM injection of V114 concomitantly with a single 0.25 mL IM injection of mRNA-1273 on Day 1, followed by a single 0.5 mL IM injection of placebo for V114 on Day 30.
  Interventions: Biological: V114; Biological: mRNA-1273; Biological: Placebo for V114
- V114 Nonconcomitant with mRNA-1273 (V114 Nonconcomitant) (Experimental): Participants received single 0.5 mL IM injection of placebo for V114 on Day 1 concomitantly with a single 0.25 mL IM injection of mRNA-1273, followed by a single 0.5 mL IM injection of V114 on Day 30.
  Interventions: Biological: V114; Biological: mRNA-1273; Biological: Placebo for V114

INTERVENTIONS:
Biological: V110 — Single intramuscular (IM) dose of 0.5 mL V110, a pneumococcal polysaccharide vaccine (PCV), containing the 23 serotypes: 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F
  Other Names: PNEUMOVAX™23; 23-Valent Pneumococcal Polysaccharide Vaccine
  Arms: V110 Concomitant with mRNA-1273 (V110 Concomitant); V110 Nonconcomitant with mRNA-1273 (V110 Nonconcomitant)
Biological: V114 — Single IM dose of 0.5 mL V114 a 15-valent PCV containing the 15 serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, 33F
  Other Names: VAXNEUVANCE™; 15-Valent Pneumococcal Conjugate; Vaccine
  Arms: V114 Concomitant with mRNA-1273 (V114 Concomitant); V114 Nonconcomitant with mRNA-1273 (V114 Nonconcomitant)
Biological: mRNA-1273 — Single IM dose of 50 μg/0.25 mL mRNA-1273
Biological: Placebo for V110 — Single IM dose of 0.5 mL placebo for V110
  Arms: V110 Concomitant with mRNA-1273 (V110 Concomitant); V110 Nonconcomitant with mRNA-1273 (V110 Nonconcomitant)
Biological: Placebo for V114 — Single IM dose of 0.5 mL placebo for V114
  Arms: V114 Concomitant with mRNA-1273 (V114 Concomitant); V114 Nonconcomitant with mRNA-1273 (V114 Nonconcomitant)

SUMMARY:
The purpose of this study is to evaluate the concomitant and non-concomitant use of messenger ribonucleic acid (mRNA) mRNA-1273, the nucleoside-modified mRNA vaccine for active immunization to prevent coronavirus disease (COVID-19) caused by severe acute respiratory syndrome coronavirus (SARS-CoV-2), with a 23-valent pneumococcal polysaccharide vaccine (V110) for the prevention of pneumococcal disease, or a 15-valent pneumococcal conjugate vaccine (V114) indicated for the prevention of invasive pneumococcal disease.

ELIGIBILITY:
Inclusion Criteria:

* Is in good health
* Any underlying chronic illness must be documented to be in stable condition
* Has received a 2-dose primary series of the Moderna mRNA SARS-CoV-2 vaccine ≥5 months before receipt of study vaccine at Visit 1
* May have received either: a) A first booster dose of the Moderna mRNA SARS-CoV-2 vaccine ≥4 months before receipt of study vaccine at Visit 1, or b) No booster dose of the Moderna mRNA SARS-CoV-2 vaccine
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a woman of childbearing potential (WOCBP) OR is a WOCBP and using an acceptable contraceptive method, or is abstinent from heterosexual intercourse

Exclusion Criteria:

* Has a current SARS-CoV-2 infection or a known history of SARS-CoV-2 infection <3 months before receipt of study vaccine at Visit 1
* Has a history of myocarditis and/or pericarditis
* Has a known or suspected impairment of immunological function including, but not limited to, a history of congenital or acquired immunodeficiency, documented human immunodeficiency virus (HIV) infection, functional or anatomic asplenia, or history of autoimmune disease
* Has a coagulation disorder contraindicating intramuscular vaccinations
* Had a recent illness with fever (defined as oral or tympanic temperature ≥100.4°F [≥38.0°C]; axillary or temporal temperature ≥99.4°F [≥37.4°C]) or received antibiotic therapy for an acute illness occurring <72 hours before receipt of study vaccine
* Has a known malignancy that is progressing or has required active treatment <3 years before receipt of study vaccine at Visit 1
* Received prior administration of a pneumococcal polysaccharide vaccine <5 years before study enrollment or is expected to receive a pneumococcal polysaccharide vaccine during the study outside the protocol
* Received prior administration of a PCV <1 year before receipt of study vaccine at Visit 1 or is expected to receive a PCV during the study outside the protocol
* Received prior administration of any SARS-CoV-2 vaccine other than the 2-dose primary series of the Moderna mRNA vaccine with or without a first booster dose, or is expected to receive any SARS-CoV-2 vaccine during the study outside the protocol
* Received prior monoclonal antibody treatment for SARS-CoV-2 infection
* Received antiviral treatment for SARS-CoV-2 infection <3 months before receipt of study vaccine at Visit 1
* Received systemic corticosteroids for ≥14 consecutive days and has not completed intervention ≥30 days before receipt of study vaccine at Visit 1
* Received systemic corticosteroids exceeding physiologic replacement doses ≤14 days before receipt of study vaccine
* Is currently receiving immunosuppressive therapy, including chemotherapeutic agents used to treat cancer or other conditions, and interventions associated with organ or bone marrow transplantation, or autoimmune disease
* Received any non-live vaccine ≤14 days before receipt of study vaccine or is scheduled to receive any non-live vaccine ≤30 days after receipt of study vaccine. Exception: Inactivated influenza vaccine allowed if given ≥7 days before or ≥15 days after receipt of study vaccine
* Received any live virus vaccine ≤30 days before receipt of study vaccine or is scheduled to receive any live virus vaccine ≤30 days after receipt of study vaccine
* Received a blood transfusion or blood products (including globulin) ≤6 months before receipt of study vaccine or is scheduled to receive a blood transfusion or blood product ≤30 days after receipt of study vaccine
* Is currently participating in or has participated in an interventional clinical study with an investigational compound or device within 2 months of participating in this current study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (46):
- United States (42):
  - Carbon Health ( Site 0045), North Hollywood, California
  - Valley Clinical Trials Inc. ( Site 0002), Northridge, California
  - Center for Clinical Trials, LLC ( Site 0022), Paramount, California
  - Artemis Institute for Clinical Research ( Site 0024), San Diego, California
  - California Research Foundation ( Site 0004), San Diego, California
  - Millennium Clinical Trials ( Site 0027), Simi Valley, California
  - Diablo Clinical Research, Inc ( Site 0043), Walnut Creek, California
  - Alliance for Multispecialty Research, LLC ( Site 0036), Coral Gables, Florida
  - Indago Research and Health Center Inc ( Site 0006), Hialeah, Florida
  - Optimal Research LLC ( Site 0019), Melbourne, Florida
  - Advanced Medical Research, LLC ( Site 0030), Miami, Florida
  - Lakes Research LLC ( Site 0012), Miami Lakes, Florida
  - Atlanta Center For Medical Research ( Site 0053), Atlanta, Georgia
  - Optimal Research ( Site 0054), Peoria, Illinois
  - Alliance for Multispecialty Research, LLC ( Site 0018), Newton, Kansas
  - AMR Lexington ( Site 0055), Lexington, Kentucky
  - Centennial Medical Group ( Site 0016), Elkridge, Maryland
  - Community Clinical Research Center ( Site 0032), Marlborough, Massachusetts
  - Alliance for Multispecialty Research, LLC ( Site 0011), Kansas City, Missouri
  - Wake Research Clinical Research Center of Nevada, LLC ( Site 0021), Las Vegas, Nevada
  - AXCES Research Group ( Site 0017), Santa Fe, New Mexico
  - Certified Research Associates ( Site 0042), Cortland, New York
  - Corning Center for Clinical Research ( Site 0052), Horseheads, New York
  - Rochester Clinical Research, Inc. ( Site 0010), Rochester, New York
  - Accellacare - Winston-Salem ( Site 0049), Winston-Salem, North Carolina
  - Velocity Clinical Research- Cleveland ( Site 0023), Cleveland, Ohio
  - Velocity Clinical Research-Providence ( Site 0015), East Greenwich, Rhode Island
  - Coastal Carolina Research Center ( Site 0044), North Charleston, South Carolina
  - Benchmark Research ( Site 0007), Austin, Texas
  - South Texas Clinical Research ( Site 0033), Corpus Christi, Texas
  - Benchmark Research ( Site 0039), Fort Worth, Texas
  - University of Texas Medical Branch at Galveston ( Site 0037), Galveston, Texas
  - Texas Center For Drug Development ( Site 0013), Houston, Texas
  - Wellness Clinical Research Associates ( Site 0051), McKinney, Texas
  - Diagnostics Research Group ( Site 0001), San Antonio, Texas
  - DM Clinical Research ( Site 0025), Tomball, Texas
  - Crossroads Clinical Research LLC ( Site 0020), Victoria, Texas
  - Velocity Clinical Research, Salt Lake City ( Site 0035), West Jordan, Utah
  - Charlottesville Medical Research Center, LLC ( Site 0008), Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc. ( Site 0014), Newport News, Virginia
  - Alliance for Multispecialty Research LLC (AMR - Norfolk) ( Site 0057), Norfolk, Virginia
  - Clinical Research Partners, LLC. ( Site 0005), Richmond, Virginia
- Puerto Rico (4):
  - Cooperativa de Facultad Medica SANACOOP ( Site 0104), Bayamón
  - CAIMED Center - Ponce School of Medicine ( Site 0103), Ponce
  - Caparra Internal Medicine Research Center. PSC ( Site 0102), Río Grande
  - Clinical Research Puerto Rico ( Site 0105), San Juan

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Omole T, Pelayo E, Weinberg AS, Chalkias S, Endale Z, Tamms G, Sterling TM, Good L, Shekar T, Johnson M, Banniettis N, Buchwald UK, Esteves-Jaramillo A. Safety, Tolerability, and Immunogenicity of the Pneumococcal Vaccines PPSV23 or PCV15 Co-Administered with a Booster Dose of mRNA-1273 SARS-CoV-2 Vaccine in Healthy Adults >/=50 Years of Age. Vaccines (Basel). 2025 Feb 15;13(2):192. doi: 10.3390/vaccines13020192. PMID 40006738
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26095&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- V110 Nonconcomitant With mRNA-1273 (V110 Nonconcomitant): Participants received a single 0.5 mL IM injection of placebo for V110 on Day 1 concomitantly with a single 0.25 mL IM vaccination of mRNA-1273, followed by a single 0.5 mL IM vaccination of V110 on Day 30.
- V114 Concomitant With mRNA-1273 (V114 Concomitant): Participants received a single 0.5 mL IM vaccination of V114 concomitantly with a single 0.25 mL IM vaccination of mRNA-1273 on Day 1, followed by a single 0.5 mL IM injection of placebo for V114 on Day 30.
- V114 Nonconcomitant With mRNA-1273 (V114 Nonconcomitant): Participants received single 0.5 mL IM injection of placebo for V114 on Day 1 concomitantly with a single 0.25 mL IM vaccination of mRNA-1273, followed by a single 0.5 mL IM vaccination of V114 on Day 30.
Period: Overall Study
Arm/Group | V110 Concomitant With mRNA-1273 (V110 Concomitant) | V110 Nonconcomitant With mRNA-1273 (V110 Nonconcomitant) | V114 Concomitant With mRNA-1273 (V114 Concomitant) | V114 Nonconcomitant With mRNA-1273 (V114 Nonconcomitant)
Started | 214 | 212 | 214 | 210
Received Any Vaccination | 214 | 211 | 210 (One participant in the V114 Concomitant Group received two doses of mRNA-1273 in error at Visit 1 and was excluded from the safety population.) | 208
Completed | 208 | 199 | 203 | 198
Not Completed | 6 | 13 | 11 | 12
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 3 | 6 | 4 | 3
Not completed — Randomized By Mistake Without Study Treatment | 0 | 0 | 4 | 1
Not completed — Withdrawal by Subject | 3 | 7 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V110 Concomitant With mRNA-1273 (V110 Concomitant) | V110 Nonconcomitant With mRNA-1273 (V110 Nonconcomitant) | V114 Concomitant With mRNA-1273 (V114 Concomitant) | V114 Nonconcomitant With mRNA-1273 (V114 Nonconcomitant) | Total
Number analyzed (Participants) | 214 | 212 | 214 | 210 | 850
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (8.1) | 60.4 (8.4) | 60.4 (7.8) | 60.3 (8.1) | 60.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 131 | 113 | 130 | 481
  Male | 107 | 81 | 101 | 80 | 369
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 87 | 98 | 90 | 93 | 368
  Not Hispanic or Latino | 127 | 112 | 124 | 116 | 479
  Unknown or Not Reported | 0 | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 2 | 3
  Asian | 4 | 3 | 7 | 4 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 41 | 33 | 36 | 40 | 150
  White | 164 | 173 | 167 | 159 | 663
  More than one race | 5 | 3 | 3 | 5 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Injection-Site Adverse Events (AEs) Among Participants Administered V110
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs include redness, swelling, pain/tenderness, and underarm gland swelling or tenderness/lymphadenopathy at the injection site. The percentage of participants with one or more solicited injection-site AEs following any vaccination was reported.
Time Frame: Up to Day 7 After Any Vaccination (Up to Study Day 37)
Population: All randomized participants who received 1 dose of V110 concomitantly or nonconcomitantly with mRNA-1273.
Measure: Number; unit: Percentage of Participants
Arm/Group | V110 Concomitant With mRNA-1273 (V110 Concomitant) | V110 Nonconcomitant With mRNA-1273 (V110 Nonconcomitant)
Number analyzed (Participants) | 214 | 211
Percentage of Participants
  Injection site erythema | 18.7 | 14.7
  Injection site pain | 74.8 | 74.4
  Injection site swelling | 23.4 | 26.5
  Lymphadenopathy | 17.3 | 25.1

2. Primary Outcome: Percentage of Participants With Solicited Injection-Site Adverse Events Among Participants Administered V114
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs include redness, swelling, pain/tenderness, and underarm gland swelling or tenderness/lymphadenopathy at the injection site. The percentage of participants with one or more solicited injection-site AEs following any vaccination was reported.
Time Frame: Up to Day 7 After Any Vaccination (Up to Study Day 37)
Population: All randomized participants who received 1 dose of V114 concomitantly or nonconcomitantly with mRNA-1273.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 Concomitant With mRNA-1273 (V114 Concomitant) | V114 Nonconcomitant With mRNA-1273 (V114 Nonconcomitant)
Number analyzed (Participants) | 209 | 208
Percentage of Participants
  Injection site erythema | 15.3 | 16.3
  Injection site pain | 70.8 | 76.9
  Injection site swelling | 20.6 | 29.3
  Lymphadenopathy | 17.7 | 25.5

3. Primary Outcome: Percentage of Participants With Solicited Systemic AEs Among Participants Administered V110
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Systemic adverse events (AEs) include headache, tiredness/fatigue, muscle aches all over body/myalgia, joint pain/arthralgia, nausea, vomiting, and chills. The percentage of participants with solicited systemic AEs following any vaccination was reported.
Time Frame: Up to Day 7 After Any Vaccination (Up to Study Day 37)
Population: All randomized participants who received 1 dose of V110 concomitantly or nonconcomitantly with mRNA-1273.
Measure: Number; unit: Percentage of Participants
Arm/Group | V110 Concomitant With mRNA-1273 (V110 Concomitant) | V110 Nonconcomitant With mRNA-1273 (V110 Nonconcomitant)
Number analyzed (Participants) | 214 | 211
Percentage of Participants
  Arthralgia | 15.4 | 17.5
  Chills | 18.7 | 17.5
  Fatigue | 40.7 | 36.5
  Headache | 29.0 | 34.1
  Myalgia | 18.7 | 24.6
  Nausea | 10.7 | 13.3
  Vomiting | 3.7 | 2.4

4. Primary Outcome: Percentage of Participants With Solicited Systemic AEs Among Participants Administered V114
Description: as for outcome 3
Time Frame: Up to Day 7 After Any Vaccination (Up to Study Day 37)
Population: All randomized participants who received 1 dose of V114 concomitantly or nonconcomitantly with mRNA-1273. One participant in the V114 Concomitant Group received 2 doses of mRNA-1273 in error and was excluded from the safety population per statistical analysis plan.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 Concomitant With mRNA-1273 (V114 Concomitant) | V114 Nonconcomitant With mRNA-1273 (V114 Nonconcomitant)
Number analyzed (Participants) | 209 | 208
Percentage of Participants
  Arthralgia | 16.7 | 18.8
  Chills | 18.7 | 18.8
  Fatigue | 41.1 | 46.6
  Headache | 29.2 | 38.0
  Myalgia | 21.5 | 26.9
  Nausea | 10.0 | 15.4
  Vomiting | 1.4 | 2.4

5. Primary Outcome: Percentage of Participants With Vaccine-Related Serious AEs (SAEs) Among Participants Administered V110
Description: Serious adverse events (SAEs) are defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in offspring of a participant, or other important medical events. V110 vaccine-related SAEs as determined by investigator are summarized.
Time Frame: Up to Month 6
Population: All randomized participants who received 1 dose of V110 concomitantly or nonconcomitantly with mRNA-1273.
Measure: Number; unit: Percentage of Participants
Arm/Group | V110 Concomitant With mRNA-1273 (V110 Concomitant) | V110 Nonconcomitant With mRNA-1273 (V110 Nonconcomitant)
Number analyzed (Participants) | 214 | 211
Percentage of Participants | 0.0 | 0.0

6. Primary Outcome: Percentage of Participants With Vaccine-Related SAEs Among Participants Administered V114
Description: SAEs are defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in offspring of a participant, or other important medical events. V114 vaccine-related SAEs as determined by investigator are summarized.
Time Frame: Up to Month 6
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 Concomitant With mRNA-1273 (V114 Concomitant) | V114 Nonconcomitant With mRNA-1273 (V114 Nonconcomitant)
Number analyzed (Participants) | 209 | 208
Percentage of Participants | 0.0 | 0.0

7. Primary Outcome: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) in Participants Administered V110
Description: Serotype-specific OPA GMTs for 14 of the serotypes contained in V110 were determined using a multiplexed opsonophagocytic assay (MOPA) at 30 days postvaccination with V110. The within-group 95% confidence intervals (CIs) were obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: Up to 30 days postvaccination with V110 (Study Day 30 for concomitant vaccination group, and Study Day 60 for nonconcomitant vaccination group, respectively)
Population: All randomized participants who received 1 dose of V110 concomitantly or nonconcomitantly with mRNA-1273, without protocol deviations substantially affecting immunogenicity endpoint results. Overall participants analyzed were the number of participants randomized and vaccinated with available serotype data; number analyzed for each serotype is the subset of overall participants analyzed without protocol deviation and with non-missing OPA serology data for the respective serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V110 Concomitant With mRNA-1273 (V110 Concomitant) | V110 Nonconcomitant With mRNA-1273 (V110 Nonconcomitant)
Number analyzed (Participants) | 214 | 211
Titers
  Serotype 1: number analyzed (Participants) | 182 | 177
  Serotype 1 | 236.0 [177.0 to 314.6] | 235.5 [188.4 to 341.1]
  Serotype 3: number analyzed (Participants) | 167 | 164
  Serotype 3 | 174.3 [138.6 to 219.2] | 284.0 [224.1 to 359.9]
  Serotype 4: number analyzed (Participants) | 182 | 165
  Serotype 4 | 1384.5 [1110.7 to 1725.9] | 1704.4 [1370.6 to 2119.5]
  Serotype 5: number analyzed (Participants) | 189 | 181
  Serotype 5 | 423.4 [324.9 to 551.7] | 376.3 [282.6 to 501.2]
  Serotype 6B: number analyzed (Participants) | 182 | 171
  Serotype 6B | 1336.7 [1038.2 to 1721] | 1326.8 [1016.7 to 1731.4]
  Serotype 7F: number analyzed (Participants) | 184 | 174
  Serotype 7F | 2614.4 [2123.8 to 3218.4] | 2420.2 [1919.6 to 3051.3]
  Serotype 9V: number analyzed (Participants) | 185 | 174
  Serotype 9V | 1651.1 [1352.0 to 2016.4] | 1809.2 [1502.2 to 2179.0]
  Serotype 14: number analyzed (Participants) | 184 | 176
  Serotype 14 | 3048.3 [2429.0 to 3825.5] | 2618.4 [2078.8 to 3298.1]
  Serotype 18C: number analyzed (Participants) | 188 | 179
  Serotype 18C | 1592.9 [1281.0 to 1980.7] | 2033.7 [1639.6 to 2522.5]
  Serotype 19A: number analyzed (Participants) | 185 | 169
  Serotype 19A | 2135.7 [1761.7 to 2589.2] | 2626.1 [2139.6 to 3223.2]
  Serotype 19F: number analyzed (Participants) | 180 | 167
  Serotype 19F | 1379.9 [1144.4 to 1663.9] | 1532.6 [1250.5 to 1878.5]
  Serotype 22F: number analyzed (Participants) | 175 | 170
  Serotype 22F | 2023.0 [1559.4 to 2624.5] | 2178.4 [1630.9 to 2909.9]
  Serotype 23F: number analyzed (Participants) | 183 | 169
  Serotype 23F | 739.0 [559.4 to 976.3] | 839.9 [639.5 to 1103.1]
  Serotype 33F: number analyzed (Participants) | 176 | 166
  Serotype 33F | 10089.0 [7799.0 to 13051.4] | 10909.2 [8634.0 to 13783.9]

8. Primary Outcome: Serotype-specific OPA GMT in Participants Administered V114
Description: Serotype-specific OPA GMTs for 15 of the serotypes contained in V114 were determined using a MOPA at 30 days postvaccination with V114. The within-group 95% CIs were obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: Up to 30 days postvaccination with V114 (Study Day 30 for concomitant vaccination group, and Study Day 60 for nonconcomitant vaccination group, respectively)
Population: All randomized participants who received 1 dose of V114 concomitantly or nonconcomitantly with mRNA-1273, without protocol deviations substantially affecting immunogenicity endpoint results. Overall participants analyzed were the number of participants randomized and vaccinated with available serotype data; number analyzed for each serotype is the subset of overall participants analyzed without protocol deviation and with non-missing OPA serology data for the respective serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V114 Concomitant With mRNA-1273 (V114 Concomitant) | V114 Nonconcomitant With mRNA-1273 (V114 Nonconcomitant)
Number analyzed (Participants) | 210 | 208
Titers
  Serotype 1: number analyzed (Participants) | 186 | 174
  Serotype 1 | 208.3 [160.8 to 269.9] | 265.6 [203.4 to 346.7]
  Serotype 3: number analyzed (Participants) | 174 | 155
  Serotype 3 | 237.5 [197.5 to 285.6] | 338.4 [275.3 to 416.0]
  Serotype 4: number analyzed (Participants) | 181 | 176
  Serotype 4 | 1586.0 [1296.5 to 1940.2] | 1758.6 [1419.4 to 2178.8]
  Serotype 5: number analyzed (Participants) | 190 | 180
  Serotype 5 | 447.0 [341.7 to 584.8] | 505.5 [382.7 to 667.8]
  Serotype 6A: number analyzed (Participants) | 176 | 162
  Serotype 6A | 4345.3 [3490.0 to 5410.1] | 5787.1 [4468.4 to 7495.0]
  Serotype 6B: number analyzed (Participants) | 173 | 158
  Serotype 6B | 3655.5 [2939.1 to 4546.6] | 4992.9 [3896.2 to 6398.2]
  Serotype 7F: number analyzed (Participants) | 187 | 170
  Serotype 7F | 3465.7 [2858.7 to 4201.6] | 3283.0 [2664.3 to 4045.4]
  Serotype 9V: number analyzed (Participants) | 187 | 166
  Serotype 9V | 1730.3 [1432.7 to 2089.8] | 2026.6 [1651.0 to 2487.5]
  Serotype 14: number analyzed (Participants) | 186 | 177
  Serotype 14 | 2487.2 [2026.1 to 3053.2] | 2460.8 [2018.4 to 3000.3]
  Serotype 18C: number analyzed (Participants) | 187 | 171
  Serotype 18C | 3144.5 [2597.3 to 3806.8] | 3183.5 [2587.9 to 3916.2]
  Serotype 19A: number analyzed (Participants) | 173 | 162
  Serotype 19A | 3214.3 [2735.5 to 3776.9] | 4037.4 [3234.4 to 5039.8]
  Serotype 19F: number analyzed (Participants) | 182 | 164
  Serotype 19F | 1742.0 [1440.1 to 2107.2] | 1950.1 [1592.9 to 2387.4]
  Serotype 22F: number analyzed (Participants) | 175 | 156
  Serotype 22F | 2282.7 [1804.7 to 2887.3] | 2670.6 [2062.6 to 3457.9]
  Serotype 23F: number analyzed (Participants) | 181 | 169
  Serotype 23F | 2326.3 [1831.2 to 2955.2] | 2212.0 [1685.3 to 2903.3]
  Serotype 33F: number analyzed (Participants) | 175 | 166
  Serotype 33F | 6788.5 [5312.9 to 8673.9] | 9339.7 [7330.9 to 11899.0]

9. Primary Outcome: SARS-CoV-2-specific Binding Antibody (bAb) GMT in Participants Administered Either V110 or V114
Description: Sera from participants were used to measure vaccine-induced bAb responses using a validated ligand-binding assay specific to the SARS-CoV-2 Spike protein at 30 days post vaccination. The within-group 95% CIs were obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution. As prespecified by the protocol and statistical analysis plan, the V110 nonconcomitant group and V114 nonconcomitant group were combined for this analysis, as they shared the same administration for the first visit (mRNA-1273 and placebo).
Time Frame: Up to 30 days postvaccination with mRNA-1273 (Study Day 30)
Population: All randomized participants who received 1 dose of either V110 or V114 concomitantly or nonconcomitantly with mRNA-1273, without protocol deviations substantially affecting immunogenicity endpoint results and with available bAb data. As prespecified by the protocol and statistical analysis plan, the V110 nonconcomitant group and V114 nonconcomitant group were combined for this analysis, as they shared the vaccinations at the first visit (mRNA-1273 and placebo).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Combined V110/V114 Nonconcomitant: Per protocol, participants received a single 0.5 mL IM injection of placebo on Day 1 concomitantly with a single 0.25 mL IM injection of mRNA-1273.
Arm/Group | V110 Concomitant With mRNA-1273 (V110 Concomitant) | V114 Concomitant With mRNA-1273 (V114 Concomitant) | Combined V110/V114 Nonconcomitant
Number analyzed (Participants) | 197 | 196 | 382
Titers | 824118.4 [717446.4 to 946650.6] | 861746.4 [756496.4 to 981639.8] | 1102295.7 [1003694.1 to 1210583.7]

10. Secondary Outcome: Serotype-specific OPA Geometric Mean Fold Rise (GMFR) in Participants Administered V110
Description: Serotype-specific OPA for 14 of the serotypes contained in V110 was determined using a MOPA. GMFR is the geometric mean fold rise from baseline to 30 days postvaccination. The within-group 95% confidence intervals (CIs) were obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: Baseline and 30 days postvaccination with V110 (Study Day 1 and Study Day 30 for concomitant vaccination group, and Study Day 30 and Study Day 60 for nonconcomitant vaccination group, respectively)
Population: All randomized participants receiving 1 dose of V110 concomitantly or nonconcomitantly with mRNA-1273, without protocol deviations substantially affecting immunogenicity endpoint results. Overall participants analyzed were the number of participants randomized and vaccinated with available serotype data; number analyzed for each serotype is the subset of overall participants analyzed without protocol deviation and with baseline and post-vaccination OPA serology data for the respective serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V110 Concomitant With mRNA-1273 (V110 Concomitant) | V110 Nonconcomitant With mRNA-1273 (V110 Nonconcomitant)
Number analyzed (Participants) | 214 | 211
Ratio
  Serotype 1: number analyzed (Participants) | 175 | 173
  Serotype 1 | 24.8 [18.3 to 33.7] | 24.2 [17.8 to 33.0]
  Serotype 3: number analyzed (Participants) | 151 | 153
  Serotype 3 | 7.1 [5.7 to 8.9] | 11.6 [9.1 to 14.8]
  Serotype 4: number analyzed (Participants) | 169 | 154
  Serotype 4 | 12.8 [9.5 to 17.3] | 15.7 [11.5 to 21.3]
  Serotype 5: number analyzed (Participants) | 180 | 176
  Serotype 5 | 15.1 [11.5 to 19.9] | 13.8 [10.4 to 18.2]
  Serotype 6B: number analyzed (Participants) | 172 | 164
  Serotype 6B | 8.2 [6.0 to 11.2] | 8.6 [6.3 to 11.6]
  Serotype 7F: number analyzed (Participants) | 170 | 162
  Serotype 7F | 14.5 [11.0 to 19.2] | 14.8 [10.8 to 20.2]
  Serotype 9V: number analyzed (Participants) | 170 | 160
  Serotype 9V | 4.3 [3.4 to 5.4] | 5.3 [4.2 to 6.7]
  Serotype 14: number analyzed (Participants) | 168 | 168
  Serotype 14 | 6.0 [4.6 to 7.7] | 7.0 [5.3 to 9.2]
  Serotype 18C: number analyzed (Participants) | 180 | 173
  Serotype 18C | 10.2 [8.1 to 12.9] | 10.9 [8.5 to 13.9]
  Serotype 19A: number analyzed (Participants) | 174 | 161
  Serotype 19A | 7.8 [6.1 to 9.9] | 8.7 [6.7 to 11.3]
  Serotype 19F: number analyzed (Participants) | 162 | 156
  Serotype 19F | 6.9 [5.3 to 8.8] | 6.7 [5.4 to 8.4]
  Serotype 22F: number analyzed (Participants) | 146 | 150
  Serotype 22F | 25.6 [16.8 to 39.0] | 30.8 [20.1 to 47.1]
  Serotype 23F: number analyzed (Participants) | 167 | 154
  Serotype 23F | 4.7 [3.5 to 6.5] | 6.2 [4.6 to 8.5]
  Serotype 33F: number analyzed (Participants) | 165 | 156
  Serotype 33F | 12.2 [8.9 to 16.7] | 16.9 [11.7 to 24.3]

11. Secondary Outcome: Serotype-specific OPA GMFR in Participants Administered V114
Description: Serotype-specific OPA for all 15 of the serotypes contained in V114 were determined using a MOPA. GMFR is the geometric mean fold rise from baseline to 30 days postvaccination. The within-group 95% CIs were obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: Baseline and 30 days postvaccination with V114 (Study Day 1 and Study Day 30 for concomitant vaccination group, and Study Day 30 and Study Day 60 for nonconcomitant vaccination group, respectively)
Population: All randomized participants receiving 1 dose of V114 concomitantly or nonconcomitantly with mRNA-1273, without protocol deviations substantially affecting immunogenicity endpoint results. Overall participants analyzed were the number of participants randomized and vaccinated with available serotype data; number analyzed for each serotype is the subset of overall participants analyzed without protocol deviation and with baseline and post-vaccination OPA serology data for the respective serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 Concomitant With mRNA-1273 (V114 Concomitant) | V114 Nonconcomitant With mRNA-1273 (V114 Nonconcomitant)
Number analyzed (Participants) | 210 | 208
Ratio
  Serotype 1: number analyzed (Participants) | 176 | 173
  Serotype 1 | 17.3 [12.8 to 23.5] | 24.5 [17.8 to 33.6]
  Serotype 3: number analyzed (Participants) | 161 | 150
  Serotype 3 | 9.0 [7.0 to 11.5] | 14.5 [11.2 to 18.8]
  Serotype 4: number analyzed (Participants) | 164 | 164
  Serotype 4 | 13.3 [9.4 to 18.6] | 20.6 [14.8 to 28.8]
  Serotype 5: number analyzed (Participants) | 183 | 179
  Serotype 5 | 14.7 [11.2 to 19.4] | 18.7 [13.9 to 25.2]
  Serotype 6A: number analyzed (Participants) | 162 | 149
  Serotype 6A | 12.7 [9.9 to 16.4] | 23.0 [17.0 to 31.0]
  Serotype 6B: number analyzed (Participants) | 164 | 153
  Serotype 6B | 19.6 [14.0 to 27.3] | 28.4 [19.8 to 40.9]
  Serotype 7F: number analyzed (Participants) | 177 | 164
  Serotype 7F | 17.6 [12.7 to 24.3] | 14.9 [10.8 to 20.4]
  Serotype 9V: number analyzed (Participants) | 175 | 158
  Serotype 9V | 4.7 [3.7 to 5.9] | 5.2 [4.1 to 6.5]
  Serotype 14: number analyzed (Participants) | 178 | 166
  Serotype 14 | 4.8 [3.6 to 6.4] | 6.3 [4.7 to 8.3]
  Serotype 18C: number analyzed (Participants) | 177 | 167
  Serotype 18C | 16.6 [12.4 to 22.3] | 17.6 [13.5 to 22.9]
  Serotype 19A: number analyzed (Participants) | 162 | 156
  Serotype 19A | 9.5 [7.1 to 12.5] | 15.2 [11.2 to 20.7]
  Serotype 19F: number analyzed (Participants) | 168 | 155
  Serotype 19F | 8.6 [6.6 to 11.2] | 9.8 [7.5 to 12.8]
  Serotype 22F: number analyzed (Participants) | 152 | 142
  Serotype 22F | 40.7 [25.7 to 64.6] | 43.9 [27.4 to 70.2]
  Serotype 23F: number analyzed (Participants) | 163 | 154
  Serotype 23F | 13.9 [10.1 to 19.1] | 17.0 [12.1 to 23.9]
  Serotype 33F: number analyzed (Participants) | 162 | 162
  Serotype 33F | 7.9 [5.8 to 10.9] | 12.4 [8.7 to 17.7]

12. Secondary Outcome: SARS-CoV-2-specific Binding Antibody (bAb) GMFR in Participants Administered Either V110 or V114
Description: Sera from participants was used to measure vaccine-induced bAb responses using a validated ligand-binding assay specific to the SARS-CoV-2 Spike protein. GMFR is the geometric mean fold rise from baseline to 30 days postvaccination. The within-group 95% CIs were obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution. As prespecified by the protocol and statistical analysis plan, the V110 nonconcomitant group and V114 nonconcomitant group were combined for this analysis, as they shared the same administration for the first visit (mRNA-1273 and placebo).
Time Frame: Baseline and 30 days postvaccination with mRNA-1273 (Study Day 1 and Study Day 30, respectively)
Population: All randomized participants who received 1 dose of either V110 or V114 concomitantly or nonconcomitantly with mRNA-1273, without protocol deviations substantially affecting immunogenicity endpoint results and with available baseline and post-vaccination bAb data. As prespecified by the protocol and statistical analysis plan, the V110 nonconcomitant group and V114 nonconcomitant group were combined for this analysis, as they shared the same vaccinations at the first visit (mRNA-1273 and placebo).
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- Combined V110/V114 Nonconcomitant: Participants received single 0.5 mL IM injection of placebo on Day 1 concomitantly with a single 0.25 mL IM injection of mRNA-1273.
Arm/Group | V110 Concomitant With mRNA-1273 (V110 Concomitant) | V114 Concomitant With mRNA-1273 (V114 Concomitant) | Combined V110/V114 Nonconcomitant
Number analyzed (Participants) | 196 | 195 | 379
Ratio | 8.6 [6.7 to 11.0] | 8.1 [6.4 to 10.2] | 9.1 [7.7 to 10.8]

13. Secondary Outcome: Percentage of Participants Who Achieve a ≥4-fold Rise in Serotype-specific OPA Responses From Baseline to 30 Days Postvaccination With V110
Description: Serotype-specific OPA for 14 of the serotypes contained in V110 was determined using a MOPA. The percentage of participants who achieved a ≥4-fold rise in OPA titer from baseline to 30 days postvaccination were calculated. The within-group 95% CIs are based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V110 Concomitant With mRNA-1273 (V110 Concomitant) | V110 Nonconcomitant With mRNA-1273 (V110 Nonconcomitant)
Number analyzed (Participants) | 214 | 211
Percentage of Participants
  Serotype 1: number analyzed (Participants) | 175 | 173
  Serotype 1 | 76.0 [69.0 to 82.1] | 75.1 [68.0 to 81.4]
  Serotype 3: number analyzed (Participants) | 151 | 153
  Serotype 3 | 66.9 [58.8 to 74.3] | 72.5 [64.8 to 79.4]
  Serotype 4: number analyzed (Participants) | 169 | 154
  Serotype 4 | 66.3 [58.6 to 73.4] | 68.2 [60.2 to 75.4]
  Serotype 5: number analyzed (Participants) | 180 | 176
  Serotype 5 | 75.0 [68.0 to 81.1] | 69.9 [62.5 to 76.6]
  Serotype 6B: number analyzed (Participants) | 172 | 164
  Serotype 6B | 55.8 [48.1 to 63.4] | 56.7 [48.8 to 64.4]
  Serotype 7F: number analyzed (Participants) | 170 | 162
  Serotype 7F | 71.2 [63.7 to 77.9] | 66.7 [58.8 to 73.9]
  Serotype 9V: number analyzed (Participants) | 170 | 160
  Serotype 9V | 47.1 [39.4 to 54.9] | 51.9 [43.8 to 59.8]
  Serotype 14: number analyzed (Participants) | 168 | 168
  Serotype 14 | 49.4 [41.6 to 57.2] | 52.4 [44.5 to 60.1]
  Serotype 18C: number analyzed (Participants) | 180 | 173
  Serotype 18C | 66.7 [59.3 to 73.5] | 69.9 [62.5 to 76.7]
  Serotype 19A: number analyzed (Participants) | 174 | 161
  Serotype 19A | 61.5 [53.8 to 68.8] | 62.1 [54.1 to 69.6]
  Serotype 19F: number analyzed (Participants) | 162 | 156
  Serotype 19F | 62.3 [54.4 to 69.8] | 60.3 [52.1 to 68.0]
  Serotype 22F: number analyzed (Participants) | 146 | 150
  Serotype 22F | 68.5 [60.3 to 75.9] | 66.0 [57.8 to 73.5]
  Serotype 23F: number analyzed (Participants) | 167 | 154
  Serotype 23F | 44.3 [36.6 to 52.2] | 53.9 [45.7 to 61.9]
  Serotype 33F: number analyzed (Participants) | 165 | 156
  Serotype 33F | 67.3 [53.5 to 74.4] | 67.9 [60.0 to 75.2]

14. Secondary Outcome: Percentage of Participants Who Achieve a ≥4-fold Rise in Serotype-specific OPA Responses From Baseline to 30 Days Postvaccination With V114
Description: Serotype-specific OPA for all 15 of the serotypes in V114 were determined using a MOPA. The percentage of participants who achieved a ≥4-fold rise in OPA titer from baseline to 30 days postvaccination were calculated. The within-group 95% CIs are based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 Concomitant With mRNA-1273 (V114 Concomitant) | V114 Nonconcomitant With mRNA-1273 (V114 Nonconcomitant)
Number analyzed (Participants) | 210 | 208
Percentage of Participants
  Serotype 1: number analyzed (Participants) | 176 | 173
  Serotype 1 | 72.7 [65.5 to 79.2] | 73.4 [66.2 to 79.8]
  Serotype 3: number analyzed (Participants) | 161 | 150
  Serotype 3 | 65.2 [57.3 to 72.5] | 79.3 [72.0 to 85.5]
  Serotype 4: number analyzed (Participants) | 164 | 164
  Serotype 4 | 68.9 [61.2 to 75.9] | 73.2 [65.7 to 79.8]
  Serotype 5: number analyzed (Participants) | 183 | 179
  Serotype 5 | 70.5 [63.3 to 77.0] | 73.2 [66.1 to 79.5]
  Serotype 6A: number analyzed (Participants) | 162 | 149
  Serotype 6A | 75.9 [68.6 to 82.3] | 82.6 [75.5 to 88.3]
  Serotype 6B: number analyzed (Participants) | 164 | 153
  Serotype 6B | 75.6 [68.3 to 82.0] | 76.5 [68.9 to 82.9]
  Serotype 7F: number analyzed (Participants) | 177 | 164
  Serotype 7F | 67.8 [60.4 to 74.6] | 65.2 [57.4 to 72.5]
  Serotype 9V: number analyzed (Participants) | 175 | 158
  Serotype 9V | 48.6 [41.0 to 56.2] | 53.2 [45.1 to 61.1]
  Serotype 14: number analyzed (Participants) | 178 | 166
  Serotype 14 | 45.5 [38.0 to 53.1] | 51.8 [43.9 to 59.6]
  Serotype 18C: number analyzed (Participants) | 177 | 167
  Serotype 18C | 72.9 [65.7 to 79.3] | 75.4 [68.2 to 81.8]
  Serotype 19A: number analyzed (Participants) | 162 | 156
  Serotype 19A | 63.6 [55.7 to 71.0] | 68.6 [60.7 to 75.8]
  Serotype 19F: number analyzed (Participants) | 168 | 155
  Serotype 19F | 66.1 [58.4 to 73.2] | 67.7 [59.8 to 75.0]
  Serotype 22F: number analyzed (Participants) | 152 | 142
  Serotype 22F | 69.1 [61.1 to 76.3] | 72.5 [64.4 to 79.7]
  Serotype 23F: number analyzed (Participants) | 163 | 154
  Serotype 23F | 65.0 [57.2 to 72.3] | 70.1 [62.2 to 77.2]
  Serotype 33F: number analyzed (Participants) | 162 | 162
  Serotype 33F | 56.2 [48.2 to 63.9] | 63.6 [55.7 to 71.0]

15. Secondary Outcome: Percentage of Participants With ≥4 Fold Rise From Baseline in SARS-CoV-2-specific bAb Response
Description: Sera from participants was used to measure vaccine-induced bAb responses using a validated ligand-binding assay specific to the SARS-CoV-2 Spike protein. The percentage of participants who achieved a ≥4-fold rise in bAb titer from baseline to 30 days postvaccination were calculated. The within-group 95% CIs are based on the exact binomial method proposed by Clopper and Pearson. As prespecified by the protocol and statistical analysis plan, the V110 nonconcomitant group and V114 nonconcomitant group were combined for this analysis, as they shared the same administration for the first visit (mRNA-1273 and placebo).
Time Frame: Baseline and 30 days postvaccination with mRNA-1273 (Study Day 1 and Study Day 30, respectively)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V110 Concomitant With mRNA-1273 (V110 Concomitant) | V114 Concomitant With mRNA-1273 (V114 Concomitant) | Combined V110/V114 Nonconcomitant
Number analyzed (Participants) | 196 | 195 | 379
Percentage of Participants | 55.1 [47.9 to 62.2] | 52.3 [45.1 to 59.5] | 55.9 [50.8 to 61.0]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were collected up to 28 days following any vaccination. Serious adverse events and all-cause mortality were reported throughout the duration of the study, up to 6 months.
Description: All-Cause Mortality reported for all randomized participants. All randomized participants who received at least 1 dose of any study vaccination and had follow-up data are analyzed in Serious Adverse Events and Other Adverse Events. One participant in the V114 Concomitant Group received two doses of mRNA-1273 in error at Visit 1 and was excluded from the safety population per statistical analysis plan.
Arm/Group | V110 Concomitant With mRNA-1273 (V110 Concomitant) | V110 Nonconcomitant With mRNA-1273 (V110 Nonconcomitant) | V114 Concomitant With mRNA-1273 (V114 Concomitant) | V114 Nonconcomitant With mRNA-1273 (V114 Nonconcomitant)
All-Cause Mortality (participants affected / at risk) | 0/214 | 0/212 | 0/214 | 1/210
Serious Adverse Events (participants affected / at risk) | 2/214 | 2/211 | 6/209 | 4/208
Other Adverse Events (participants affected / at risk) | 171/214 | 170/211 | 163/209 | 172/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V110 Concomitant With mRNA-1273 (V110 Concomitant) (N=214) | V110 Nonconcomitant With mRNA-1273 (V110 Nonconcomitant) (N=211) | V114 Concomitant With mRNA-1273 (V114 Concomitant) (N=209) | V114 Nonconcomitant With mRNA-1273 (V114 Nonconcomitant) (N=208)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V110 Concomitant With mRNA-1273 (V110 Concomitant) (N=214) | V110 Nonconcomitant With mRNA-1273 (V110 Nonconcomitant) (N=211) | V114 Concomitant With mRNA-1273 (V114 Concomitant) (N=209) | V114 Nonconcomitant With mRNA-1273 (V114 Nonconcomitant) (N=208)
Lymphadenopathy (Blood and lymphatic system disorders) | 37 (37) | 53 (53) | 37 (37) | 53 (54)
Nausea (Gastrointestinal disorders) | 23 (23) | 28 (28) | 22 (22) | 32 (32)
Chills (General disorders) | 40 (40) | 37 (37) | 40 (40) | 39 (39)
Fatigue (General disorders) | 88 (89) | 78 (78) | 86 (87) | 99 (100)
Injection site erythema (General disorders) | 40 (40) | 31 (31) | 32 (32) | 36 (36)
Injection site pain (General disorders) | 160 (160) | 157 (158) | 148 (148) | 160 (161)
Injection site swelling (General disorders) | 50 (50) | 56 (56) | 43 (43) | 61 (61)
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 (33) | 37 (38) | 35 (35) | 40 (40)
Myalgia (Musculoskeletal and connective tissue disorders) | 41 (41) | 53 (55) | 45 (45) | 56 (56)
Headache (Nervous system disorders) | 65 (67) | 72 (75) | 62 (65) | 79 (81)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. A coordinating investigator will be designated by mutual agreement. If publication activity is not directed by Sponsor, investigator agrees to submit all manuscripts or abstracts to Sponsor before submission, allowing Sponsor to protect proprietary information and provide comments. Authorship will be determined by mutual agreement in line with ICMJE authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT05158140/Prot_SAP_000.pdf